CLINICAL TRIAL: NCT03853447
Title: Characterization of Fibro-inflammation During Progression From Acute to Chronic Pancreatitis
Brief Title: Fibro-inflammatory Progression From Acute to Chronic Pancreatitis
Status: Recruiting | Type: Observational
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Lise Gluud, Associate Professor, Copenhagen University Hospital, Hvidovre
Other Study IDs: H-18017281
Record Dates: First submitted 2019-02-14; First posted 2019-02-25 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Pancreatitis; Acute Pancreatitis; Recurrent Pancreatitis; Chronic Pancreatitis; Inflammation; Fibrosis
MeSH Terms: conditions — Pancreatitis; Pancreatitis, Chronic; Inflammation; Fibrosis | interventions — Diagnostic Imaging; Magnetic Resonance Imaging; Endosonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum and buffy coat
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diagnostic imaging: The progression of fibrosis will be assessed based on diagnostic imaging of thre subgroups including
  Patients with chronic pancreatitis (CP; N=50) of any aetiology, except gallstones, based on MANNHEIM.
  Patients with their first attack of acute pancreatitis (AP; N=50) of any aetiology except gallstones using the revised Atlanta criteria for AP.
  Patients with recurrent AP (RAP; N=50) except gallstones, defined as two or more cases of AP as diagnosed by the revised Atlanta Criteria.
  Interventions: Diagnostic Test: Diagnostic imaging

INTERVENTIONS:
Diagnostic Test: Diagnostic imaging — MRI assessments including magnetic resonance cholangiopancreatography (MRCP) and diffusion weighted imaging (DWI) combined with gold standard EUS
  Other Names: MRI and EUS

SUMMARY:
Observational prospective study evaluating the developement of chronic pancreatitis based on imaging modalities as well as biochemical markers of inflammation, fibrosis and oxidative stress.

DETAILED DESCRIPTION:
Chronic pancreatitis (CP) represents the end-stage of a continuous disease process evolving from acute pancreatitis (AP), over recurrent acute pancreatitis (RAP). Due to the irreversible nature of CP, early detection and prevention is key. The study uses state-of-the-art imaging modalities as well as biochemical markers of to evaluate fibrosis progression in patients with pancreatitis.

The included participants have either first time AP, RAP, early CP with preserved pancreatic exocrine and endocrine function or end-stage CP with exocrine insufficiency. Included patients will be followed prospectively for 15 years with advanced MRI and contrast enhanced EUS with elastography, assessment of endocrine and exocrine pancreatic function, biochemical and nutritional assessment, and evaluation of pain processing using quantitative sensory testing. Blood for a biobank will be obtained. The purpose of the biobank is to allow analyses of potential biomarkers for the progression of disease eventually leading to CP.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CP (N=50) of any aetiology except gallstone induced CP: CP will be diagnosed based on MANNHEIM criteria .
* Cohort 2: Patients with their first attack of AP of any aetiology except gallstone induced AP (N=50). The revised Atlanta criteria for acute pancreatitis will be used as diagnostic criteria.
* Cohort 3: Patients with RAP (N=50) except gallstone induced RAP. RAP is defined as two or more cases of AP as diagnosed by the revised Atlanta Criteria.

Exclusion Criteria:

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with CP, AC pr RAP who are not:
  1. Pregnant or lactating patients
  2. Contraindications to magnetic resonance imaging (MRI) or endoscopic ultrasound
  3. Known chronic liver disease, chronic renal failure, malignancy, chronic inflammatory bowel syndrome, chronic obstructive lung disease, pulmonary fibrosis.
  4. Treatment with anti-inflammatory drugs of any kind at the time of inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-02-14 (Actual); Primary Completion 2040-01-01 (Estimated); Study Completion 2041-01-01 (Estimated)

PRIMARY OUTCOMES:
Fibrosis progression on endoscopic ultrasound (EUS) or magnetic resonance imaging (MRI) | 15 years
  Progression of fibrosis in the pancreas based on either EUS or MRI

SECONDARY OUTCOMES:
Lean body mass assessed using bioimpedance | 15 years
  Body composition focusing on lean body mass will be assessed using bioimpedance

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Gastrounit, Copenhagen University Hospital Hvidovre, Hvidovre, Capital Region Denmark
  - Department of Gastroenterology & Hepatology, Aalborg University Hospital, Aalborg
  - Abdominal Centre, Bispebjerg University Hospital, Copenhagen

IPD SHARING:
Plan to Share IPD: No